CLINICAL TRIAL: NCT03274739
Title: Maternal Mediterranean Diet During Pregnancy in Association to Longitudinal Body Mass Index Trajectories and Cardiometabolic Risk in Early Childhood
Brief Title: Maternal Diet, Body Mass Index Trajectories and Cardiometabolic Risk in Early Childhood
Status: Completed | Type: Observational
Sponsor: Barcelona Institute for Global Health (Other)
Responsible Party: Principal Investigator, Jordi Virgili, Quality Manager, Barcelona Institute for Global Health
Other Study IDs: Creal
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Cardiometabolic Risk; Growth; Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women

SUMMARY:
This study focused on evaluating the association between adherence to the Mediterranean diet during pregnancy and offspring longitudinal body mass index trajectories and cardiometabolic risk in early-childhood. This study is part of a secondary data analysis of the INMA (INfancia y Medio Ambiente-(Environment and Childhood)) Project.

ELIGIBILITY:
Inclusion Criteria:

* to be resident in one of the study areas
* to be at least 16 years old
* to have a singleton pregnancy
* to wish to deliver in the reference hospital

Exclusion Criteria:

* to not be fluent in Spanish or other regional languages.
* to have followed a programme of assisted reproduction

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study included pregnant women recruited between 2003 and 2008 in the four Spanish regions of Asturias, Gipuzkoa, Sabadell and Valencia as part of the population-based INMA ("INfancia y Medio Ambiente") birth cohort study. The pregnant women were recruited during prenatal visits in the 1st trimester of pregnancy at public health care centers or hospitals. Mothers were afterwards followed at 3rd trimester, and their children later, and at ages 6 months, 1 and 4 years.
Sampling Method: Non-Probability Sample
Enrollment: 2762 (Actual)
Dates: Start 2004-02 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2017-01-18 (Actual)

PRIMARY OUTCOMES:
Offspring's body mass index z-score trajectories | From birth to 4 years of age
Child cardiometabolic risk score | At 4 years

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guxens M, Ballester F, Espada M, Fernandez MF, Grimalt JO, Ibarluzea J, Olea N, Rebagliato M, Tardon A, Torrent M, Vioque J, Vrijheid M, Sunyer J; INMA Project. Cohort Profile: the INMA--INfancia y Medio Ambiente--(Environment and Childhood) Project. Int J Epidemiol. 2012 Aug;41(4):930-40. doi: 10.1093/ije/dyr054. Epub 2011 Apr 5. No abstract available. PMID 21471022